CLINICAL TRIAL: NCT06987006
Title: Effects of Education With Jigsaw Technique on Diabetic Foot Risk Knowledge and Self-Efficacy in Nursing Students: A Randomized Controlled Trial
Brief Title: Effects of Education With Jigsaw Technique on Diabetic Foot Risk Knowledge and Self-Efficacy in Nursing Students
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Çankırı Karatekin University (Other)
Responsible Party: Principal Investigator, Asli Tok Ozen, Assistant Professor, Çankırı Karatekin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CKU-NURSING-ATO-01
Record Dates: First submitted 2025-05-13; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Nursing Education
Keywords: Jigsaw Technique; Diabetic foot assessment; Self-efficacy

STUDY DESIGN:
Intervention Model Description: Participants included in the study will be assigned to Jigsaw education group and classical education groups in accordance with the randomized controlled study plan design. Education will be given to Jigsaw education group using the jigsaw technique. And education will be given to the classical education group using the classical education technique. Then, the diabetic foot risk knowledge level and self-efficacy of the students will be evaluated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Jigsaw Education Group (Experimental): The education will be given to this group with jigsaw education technique
  Interventions: Other: Jigsaw education
- Classical Education Group (Experimental): The education will be given to this group with classical education by instructor
  Interventions: Other: Classical Education Technique

INTERVENTIONS:
Other: Jigsaw education — The Jigsaw Technique (JT) is used as a teaching technique where each student creates pieces of an academic and instructional puzzle, specializes in puzzle groups, and teaches the subject they specialize in to other group members.
  Arms: Jigsaw Education Group
Other: Classical Education Technique — In the classical education method, students listen to the lesson explained by the educator in a classroom environment.
  Arms: Classical Education Group

SUMMARY:
The aim of this study is to evaluate the effects of education given with the jigsaw technique on the diabetic foot risk knowledge and self-efficacy in nursing students

DETAILED DESCRIPTION:
One of the important roles of nurses, the 'educational role', aims to provide the necessary behaviors for the protection, development and maintenance of health through planned education given by the nurse to healthy/sick individuals and their relatives. The focus of patient education is to provide the individual with self-management through skill and behavioral change. The provision of knowledge and skills to nurses to fulfill the requirements of the educational role begins during the student period and continues. The development of knowledge and skills for the assessment of diabetic foot risk will affect the quality of care that nursing students will provide to their patients when they start their profession after graduation. In recent years, methods and tools that facilitate learning and positively affect learning outcomes have been frequently used in education processes in order to strengthen nursing education and train more equipped nurses before graduation. One of these methods, the jigsaw (collaborative learning) model, is used to improve learning outcomes. The Jigsaw Technique (JT) is used as a teaching technique in which each student creates pieces of an academic and educational puzzle, specializes in puzzle groups and teaches the subject they specialize in to other group members. When the literature is examined, there are a limited number of studies on the jigsaw technique in the education of health professionals and students, and no study showing its effect on diabetic foot risk assessment was found.

ELIGIBILITY:
Inclusion Criteria:

* Agree to participate in the study

Exclusion Criteria:

* Don't agree to participate in the study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-06-10 (Estimated); Primary Completion 2025-06-20 (Estimated); Study Completion 2025-06-20 (Estimated)

PRIMARY OUTCOMES:
Change in knowledge level of diabetic foot risk | 1 weeks
  After the education, the difference in the knowledge level of the students regarding determining diabetic foot risk will be evaluated. The students will be given an exam that includes diabetic foot risks, signs and symptoms, and evaluation methods.
Change in self-efficacy level | 1 weeks
  The change in students' self-efficacy levels will be evaluated before and after the education. For this purpose, a student self-assessment scale with validity and reliability will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Aslı Tok Özen, Assis. Prof., Study Director — Çankırı Karatekin Universitesi
Locations (1):
- Çankırı Karatekin University, Çankırı, Çankırı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No